CLINICAL TRIAL: NCT03279887
Title: Usefulness of Lung Ultrasonography for Diagnosis of Pneumonia After Major Cardiac Surgery: a Pilot Study
Brief Title: Lung Ultrasonography After Major Cardiac Surgery
Acronym: ECHOVAP
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Adrien Bouglé, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: ECHOVAP
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pneumonia; Cardio/Pulm: Respiratory Failure; Cardiopulmonary Bypass
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post operative respiratory failure: Patients with acute respiratory failure (ARF) less than 72 hours after a major cardiac surgery with cardiopulmonary bypass
  ARF was defined as one of the following conditions:
  * If mechanical ventilation, a partial pressure of oxygen/ inspired oxygen fraction ratio (PaO2/FiO2) < 200, or failure of weaning (failure of spontaneous ventilation test, re-intubation in the first 24 hours), or need for non-invasive ventilation immediately after extubation,
  * If spontaneous ventilation: clinical signs of acute respiratory distress (dyspnea at least exertion, cyanosis, polypnea> 25/min, upper or intercostal swallowing, abdominal swing ...), pulse oximetry (SpO2) < 90% or PaO2 <60 mmHg despite oxygen therapy ≥ 3 L/min.
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound

SUMMARY:
Diagnosis of pneumonia remains difficult in intensive care unit (ICU), notably after cardiac surgery. Lung ultrasonography (LUS) has been successfully used for diagnosis of pneumonia, but its usefulness and reliability was never evaluated after cardiac surgery. This study investigates the clinical relevance of LUS for pneumonia diagnoses in cardiac ICU.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with sternotomy and cardio-pulmonary bypass (CPB) less than 3 days before
* At least one component suggestive of ARF:

  * If mechanical ventilation, a PaO2 / FiO2 ratio <200, or failure of weaning (failure of spontaneous ventilation test, re-intubation in the first 24 hours), or need for non-invasive ventilation immediately after extubation,
  * If spontaneous ventilation: clinical signs of acute respiratory distress (dyspnea at least exertion, cyanosis, polypnea> 25/min, upper or intercostal swallowing, abdominal swing ...), SpO2 < 90% or PaO2 <60 mmHg despite oxygen therapy ≥ 3L/min.

Exclusion Criteria:

* Minor patients
* Pregnancy
* Sleep apnea syndrome
* Participation refusal

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute respiratory failure after cardiac surgery and hospitalized in the surgical Intensive Care Unit of ICU of Cardiology Institute, Pitié Salpêtrière University Hospital, Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Final diagnosis of pneumonia | During the 72 hours following surgery
  Pneumonia or excluded pneumonia, was determined by consensus of 3 investigators, after an independent post hoc review of the medical records. Pneumonia diagnosis was based on concordance of clinical and radiological criteria (≥ 2 criteria including fever> 38.5 ° C or T <36 ° C, leukocytosis> 10 ^ 9 / L or leukopenia <4.10 ^ 8 / L, purulent tracheal secretions and the appearance or persistence of an infiltrate on the CXR).
  It should be confirmed by culture of a respiratory specimen: protected distal sampling with a threshold of significance ≥ 10 ^ 3 colony forming unit/mL or bronchoalveolar lavage with a threshold of significance ≥ 10 ^ 4 CFU/mL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dureau P, Bougle A, Melac AT, Ait Hamou N, Arbelot C, Ben Hassen K, Charfeddine A, Deransy R, Arcile G, Rouby JJ, Granger B, Amour J. Colour Doppler ultrasound after major cardiac surgery improves diagnostic accuracy of the pulmonary infection score in acute respiratory failure: A prospective observational study. Eur J Anaesthesiol. 2019 Sep;36(9):676-682. doi: 10.1097/EJA.0000000000001022. PMID 31107351